CLINICAL TRIAL: NCT05450783
Title: Tissue and Metabolic Characterization of Arrhythmogenic Cardiomyopathies by Hybrid PET-MRI Imaging, Impact of the Observed Profiles on the Phenotype and on the Evolution of Cardiomyopathy
Acronym: CharACTPET-MR
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Brest (Other); University Hospital, Paris (Other); University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC22_0010
Record Dates: First submitted 2022-05-16; First posted 2022-07-11 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Arrhythmogenic Cardiomyopathies
Keywords: Arrhythmogenic cardiomyopathies; PET-MR imaging; Myocardial inflammation; Prognosis; Cardiac auto-antibodies
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Patients and their relatives affected with left ventricular or biventricular AC and carrier of a pathogenic or likely pathogenic variant in one of the following genes : PKP2, DSG2, DSC2, JUP, DSP, DES, FLNC, PLN, LMNA, TMEM43, CDH2, BAG3, RYR2, RBM20
  Interventions: Other: Biocollection

INTERVENTIONS:
Other: Biocollection — serum

SUMMARY:
Status of the research project: The main complications of arrhythmogenic cardiomyopathies (AC) are sudden death, more rarely heart failure. Recently, data are emerging in favor of an associated role of myocardial inflammation and myocarditis in this pathology, but the impact of inflammation on the presentation and prognosis of the cardiomyopathy, as well as its mechanisms, are not clearly elucidated. To date, endomyocardial biopsy is the gold standard for documenting myocardial inflammation.

Aim of the research: To evaluate the interest of a new hybrid PET-MR imaging tool for tissue and metabolic characterization of AC associating MRI and 18F-FDG PET, already used in inflammatory pathologies (cardiac sarcoidosis).

Project description: Multicentric observational study of 80 patients with genetic AC undergoing PET-MR. Description of the observed profiles and their impact on the phenotype of the cardiomyopathy and its evolution, study of associated immunological mechanisms, correlation with available anatomopathological data.

Expected results and perspectives: first non-invasive description of tissue and metabolic phenotype of AC by PET-MR imaging and its prognostic role, basis for pathophysiological and therapeutic research in case of confirmation of the performances of this imaging for the detection of myocardial inflammation.

DETAILED DESCRIPTION:
Status of the research project: The main complications of arrhythmogenic cardiomyopathies (AC) are sudden death, more rarely heart failure. Recently, data are emerging in favor of an associated role of myocardial inflammation and myocarditis in this pathology, but the impact of inflammation on the presentation and prognosis of the cardiomyopathy, as well as its mechanisms, are not clearly elucidated. To date, endomyocardial biopsy is the gold standard for documenting myocardial inflammation.

Aim of the research: To evaluate the interest of a new hybrid PET-MR imaging tool for tissue and metabolic characterization of AC associating MRI and 18F-FDG PET, already used in inflammatory pathologies (cardiac sarcoidosis).

Project description: Multicentric observational study of 80 patients with genetic AC undergoing PET-MR. Description of the observed profiles and their impact on the phenotype of the cardiomyopathy and its evolution, study of associated immunological mechanisms, correlation with available anatomopathological data.

Expected results and perspectives: first non-invasive description of tissue and metabolic phenotype of AC by PET-MR imaging and its prognostic role, basis for pathophysiological and therapeutic research in case of confirmation of the performances of this imaging for the detection of myocardial inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female over 16 years old

Exclusion Criteria:

* Patients and their relatives with left ventricular or biventricular AC and carrier of a pathogenic or likely pathogenic variant in one of the following genes : PKP2, DSG2, DSC2, JUP, DSP, DES, FLNC, PLN, LMNA, TMEM43, CDH2, BAG3, RYR2, RBM20 Consent form

Exclusion Criteria :

* Sarcoidosis or known or diagnosed autoimmune disease
* History of myocardial infarction
* Patient under guardianship, curatorship or safeguard of justice

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients and their relatives with left ventricular or biventricular AC and carrier of a pathogenic or likely pathogenic variant in one of the following genes : PKP2, DSG2, DSC2, JUP, DSP, DES, FLNC, PLN, LMNA, TMEM43, CDH2, BAG3, RYR2, RBM20
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PET-RMI patients profile | one hour
  Rate of patients observed in the different expected PET-MRI patterns in the left ventricle (no late enhancement and no PET fixation, late enhancement and no PET fixation, concordant late enhancement and PET fixation, discordant late enhancement and PET fixation).

SECONDARY OUTCOMES:
PET-RMI patterns in the right ventricle | one hour
  Rate of patients with different expected PET-MRI patterns in the right ventricle (no late enhancement and no PET fixation, late enhancement and no PET fixation, concordant late enhancement and PET fixation, discordant late enhancement and PET fixation)
Prognosis according to PET-RMI patterns | 15-32 months
  Comparison of event rates (death, heart transplantation, resuscitated sudden death, hemodynamically unstable VT, syncopal VT, hospitalization for heart failure, myocarditis) observed during follow-up according to the different expected LV and RV PET-MRI profiles observed at inclusion
Cardiac auto-antibodies according to PET-RMI patterns | one hour
  Comparison of the rates of patients with circulating cardiac autoantibodies detected by indirect immunofluorescence technique according to the different expected LV and RV PET-MRI profiles at inclusion
Spatial concordance | one hour
  Rate of spatial concordance of segments with late enhancement and PET fixation on bulls-eye representations according to AHA segmentation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Piriou, PH, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CHU de Nantes, Nantes
  - AP-HP La Salpêtrière, Paris
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No